CLINICAL TRIAL: NCT03485586
Title: Comparison of the Visual Quality of Traditional Ultrasound Biometrics and Lenstar on the Cataract After Pars Plana Vitrectomy
Acronym: PPV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bojie Hu (Other)
Responsible Party: Sponsor-Investigator, Bojie Hu, Bojie Hu, Head of Ophthalmology department, Principal Investigator, Associate Senior Physician, Tianjin Medical University Eye Hospita, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Other Study IDs: HBJ 161718
Record Dates: First submitted 2018-03-24; First posted 2018-04-02 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Diabetic Retinopathy Patients After Vitrectomy
Keywords: cataract, higher order aberration,vitrectomy,diabetic retinopathy
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group:Traditional ultrasonic biological: The measurement of axial length was performed in 60 eyes (30 eyes for each group) with senile cataract of vitrectomised eye of diabetic retinopathy using lenstar and traditional ultrasonic biological combined with cornea curvimeter.In this group,we use traditional ultrasonic biological combined with cornea curvimeter to measure the ocular parameter.
  Interventions: Device: Traditional ultrasound biometrics
- Group:Lenstar: The measurement of axial length was performed in 60 eyes (30 eyes for each group) with senile cataract of vitrectomised eye of diabetic retinopathy using lenstar and traditional ultrasonic biological combined with cornea curvimeter.In this group,we use lenstar to measure the ocular parameter.
  Interventions: Device: Lenstar

INTERVENTIONS:
Device: Traditional ultrasound biometrics — To evaluate the clinical feasibility of using a new optical coherence interferometry ( lenstar ),comparing with traditional ultrasonic biometry and keratometry in the accuracy and characteristics for intraocular lens calculation of cataract after PPV
  Groups: Group:Traditional ultrasonic biological
Device: Lenstar — To evaluate the clinical feasibility of using a new optical coherence interferometry ( lenstar ),comparing with traditional ultrasonic biometry and keratometry in the accuracy and characteristics for intraocular lens calculation of cataract after PPV
  Groups: Group:Lenstar

SUMMARY:
Comparison of the visual quality of traditional ultrasound biometrics and lenstar on the cataract patients with diabetic retinopathy after vitrectomy in the 3 months later.To evaluate the clinical value of lenstar in post-vitrectomy patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cataract after vitrectomy because of diabetic retinopathy.
2. Patients with good fixation in order to cooperate with various examination.

Exclusion Criteria:

1. Myopia of >6 diopters
2. Ocular trauma and other eye disease accepted vitrectomy,such as branch retinal vein occlusion(BRVO),central retinal vein occlusion(CRVO).
3. Vision acuity <0.1
4. Silicone oil eye

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cataract after vitrectomy because of diabetic retinopathy.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-04-03 (Estimated); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
the visual quality of the eye after surgery | one month
  the visual quality of the eye after surgery through optical path difference scan（OPD Scan）
the visual quality of the eye after surgery | three month
  the visual quality of the eye after surgery through optical path difference scan（OPD Scan）

CONTACTS AND LOCATIONS:
Overall Officials: bojie Hu, docter, Study Director — Tianjin Medical University Eye Hospital
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided